CLINICAL TRIAL: NCT06865846
Title: Treatment Hypertension to Recommended Levels in Old Patients
Acronym: THReshOld
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Collaborators: Russian Gerontological Scientific and Clinical Center (Unknown); Pirogov Russian National Research Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: THReshOld2024
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Arterial Hypertension
Keywords: arterial hypertension; remote monitoring; mHealth; telemedicine; geriatric; elderly people
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BP <135 (Experimental): Higher target BP group (less than 135 mmHg). Achievement of target BP, assessment of symptoms and frequency of hypotensive episodes will be assessed.
  Interventions: Device: TeleMedBot
- BP <125 (Experimental): Higher target BP group (less than 125 mmHg). Achievement of target BP, assessment of symptoms and frequency of hypotensive episodes will be assessed.
  Interventions: Device: TeleMedBot

INTERVENTIONS:
Device: TeleMedBot — The patient will receive a questionnaire daily containing a list of questions about blood pressure and heart rate. For this purpose, a messaging application will be installed on the patients' smartphones before the study begins. All patients will be instructed and trained to use the application. Every day at 12 noon, patients will receive a questionnaire containing 2 questions. Patients can start, pause, and continue answering for 12 hours before the next questionnaire appears. For security reasons, no personal data of patients is entered or saved in the program. The research physician will receive daily information about the patient's self-monitoring results and make decisions about the need to adjust therapy.

SUMMARY:
After checking the patient characteristics to the inclusion and exclusion criteria, and confirming the ability to complete the questionnaires provided by the study protocol, patients will be randomly assigned to 2 groups: a group with a higher target BP level (less than 135 mmHg) and a lower target BP level (less than 125 mmHg). Achievement of target BP levels will be assessed using a remote monitoring system. The study will identify factors that prevent achievement of target BP levels, as well as assess the efficacy, safety and tolerability of antihypertensive therapy (AHT).

DETAILED DESCRIPTION:
The study duration is 3 months. It is planned to include at least 60 patients in the study. Before any procedures related to the study, the patient must be provided with comprehensive information about the study product, possible risks associated with its use and / or participation in the study. The study participant must provide written consent to participate in the study. At the first face-to-face visit, informed voluntary consent will be obtained in both groups, a physical examination will be performed, including measuring blood pressure, heart rate, and an orthostatic test. Monitoring will be based on measurements of office blood pressure by a doctor at the stage of inclusion in the study, as well as by the patient himself during home blood pressure measurements daily for 3 months and after 3 months at a follow-up visit to the doctor. BP will be measured with an automatic/semiautomatic tonometer in a sitting position after at least 5 minutes of rest, twice on the right and left arms, then BP will be measured on the arm with the higher systolic BP level, first in a horizontal position, then the patient will be asked to stand up and BP will be measured 45 seconds, 3 and 6 minutes after moving to a vertical position. HR will be assessed with the patient in a sitting position, lying down and 45 seconds, 3 and 6 minutes after moving to orthostasis. For the orthostatic test, the results of BP measurements while lying down and 1, 3 and 6 minutes after moving to orthostasis will be used. Orthostatic hypotension will be diagnosed with a decrease in systolic BP by 20 mmHg or more or diastolic BP by 10 mmHg or more, or a decrease in both parameters. Patients will be taught the rules for measuring BP at home. Specialized questionnaires will be filled in, combined antihypertensive therapy will be prescribed according to clinical guidelines. Daily contact using remote access: blood pressure control during home measurement and remote monitoring in case of an episode of arterial hypotension, symptom assessment using an additional questionnaire in the chatbot, and therapy adjustment if necessary.

Main objective: During the implementation of an open randomized clinical trial using home blood pressure (BP) measurement data and a remote monitoring system (TeleMedBot) for the efficacy and safety of AHT therapy, to test the hypothesis that achieving lower recommended target BP levels will be no less safe than achieving higher recommended target BP levels in elderly and senile patients with hypertension.

Optimization of drug therapy will be carried out by the research physician throughout the study.

Weekly throughout the study, the patient will be contacted to assess the safety of drug therapy and decide on AHT optimization.

The patient will also have a chatbot installed on their electronic device. The patient will be trained to work with it and will be able to ask all the questions they are interested in related to its operation. The questionnaire will consist of 2 questions and will be sent twice a day at 12:00 and 21:00. It is recommended to fill it out every day. When signs of a decrease in blood pressure are detected, the patient will be asked to fill out an additional questionnaire on the tolerability of therapy and additional telephone contact will be established with them to determine further tactics.

The patient will be explained that this chatbot is intended for systematic monitoring of health indicators and cannot respond to emergency conditions and, moreover, in no case can it replace a physical visit to a clinic, another medical institution or calling an ambulance. Therefore, the patient will be explained that if such situations arise, they should immediately contact a medical institution or call an ambulance and not rely on this platform.

After 3 months, the patient will be invited for a follow-up visit using telemedicine technologies. On this day, a follow-up survey will be conducted, the doctor will perform a physical examination of the patient, the therapy taken, and give recommendations on further treatment tactics.

TeleMedBot does not store the patient's personal data. Each patient participating in remote monitoring is coded, only the research doctor has access to personal data.

Statistical data processing is expected to be performed using IBM ® SPSS ® Statistics version 23.0 (SPSS Inc., USA). Quantitative variables will be presented as M±SD, where M is the mean and SD is the standard deviation. For clarity, ordinal variables will be presented simultaneously as Me (25%; 75%), where Me is the median, 25% and 75% are the 25th and 75th percentiles, and as M±SD. For qualitative and categorical variables (gender, anamnesis data, frequency of deviations according to physical examination data, etc.), the number and proportion of patients will be indicated. For intergroup comparisons, the Kruskal-Wallis test (for quantitative and ordinal variables) and Pearson's χ2 or two-sided Fisher's exact test (for qualitative variables) were used. Differences with a two-sided p value <0.05 will be considered statistically significant. Comparisons between groups will be made using Win ratio analysis using a hierarchical approach to the visualized indicators (see evaluation criteria).

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 65 years and older with hypertension previously diagnosed based on repeated measurements in a medical institution.

Exclusion Criteria:

1. Diagnosed dementia or severe cognitive impairment.
2. Inability to fill in questionnaires specified in the study protocol.
3. Inability to use automatic devices for recording blood pressure at home.
4. Inability to use electronic devices required for remote monitoring of home blood pressure measurements and patient well-being.
5. Presence of hemodynamically significant valvular heart defects.
6. Presence of severe renal impairment (eGFR <30 ml/min/1.73 m2) and/or increased blood creatinine levels to 221 μmol
7. Myocardial infarction or stroke within the previous 6 months.
8. Chronic heart failure with EF ≤ 40%.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Achievement of recommended target BP level | 1 month
  Achievement of recommended target BP level

SECONDARY OUTCOMES:
Assessment of the frequency of hypotensive episodes and the occurrence of hypotensive symptoms | 3 months
  Assessment of the frequency of hypotensive episodes and the occurrence of hypotensive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Gilyarevskiy, PhD, Principal Investigator — Pirogov Russian National Research Medical University
Locations (1):
- I.M. Sechenov First Moscow State Medical University of the Ministry of Health of the Russian Federation (Sechenov University), University Clinical Hospital No.1, Russian Gerontological Scientific and Clinical Center, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
According to the Local Ethics Committee rules, we are not allowed to provide this data.